CLINICAL TRIAL: NCT00863525
Title: A Double-Blind, Randomized, 2-Period Crossover, Placebo Controlled Study to Asses the Effects of a Light Breakfast on the Safety, Tolerability, and Pharmacokinetics of Single Oral Dose of MK0822
Brief Title: A Study to Assess the Effects of a Light Breakfast on the Safety, Tolerability, and Pharmacokinetics of Odanacatib (MK0822)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-006; 2009_563
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Odanacatib
  Interventions: Drug: odanacatib
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: odanacatib — A single oral dose of 100 mg odanacatib administered with a light meal in one treatment period and without a meal in the other treatment period. There will be 10 days between treatment periods.
  Other Names: MK0822
  Arms: 1
Drug: Comparator: Placebo — A single oral dose of Placebo to odanacatib administered with a light meal in one treatment period and without a meal in the other treatment period. There will be 10 days between treatment periods.
  Arms: 2

SUMMARY:
This study will assess the safety and tolerability of single doses of odanacatib (MK0822) when administered with a light breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male and between the ages of 18 and 45
* Subject is within 25% of ideal body weight and weighs between 55 and 95 kg
* Subject is in generally good health
* Subject is a nonsmoker

Exclusion Criteria:

* Subject has multiple or severe allergies to food or medications
* Subject has a history of metabolic bone disease, kidney/bladder stones, or treatment with bisphosphonates
* Subject has any infections, including HIV
* Subject has donated blood or taken another investigational drug in the last month
* Subject consumes excessive amounts of caffeine or alcohol
* Subject has a history of any illness that may confound the results of the study or pose additional risk in administering the study drug

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2004-11; Primary Completion 2004-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MK0822 based on clinical and laboratory adverse experiences | Throughout the study
Effect of a low-fat meal on pharmacokinetics of MK0822 | Through 240 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Stoch SA, Zajic S, Stone JA, Miller DL, van Bortel L, Lasseter KC, Pramanik B, Cilissen C, Liu Q, Liu L, Scott BB, Panebianco D, Ding Y, Gottesdiener K, Wagner JA. Odanacatib, a selective cathepsin K inhibitor to treat osteoporosis: safety, tolerability, pharmacokinetics and pharmacodynamics--results from single oral dose studies in healthy volunteers. Br J Clin Pharmacol. 2013 May;75(5):1240-54. doi: 10.1111/j.1365-2125.2012.04471.x. PMID 23013236